CLINICAL TRIAL: NCT07198061
Title: Efficacy and Safety of Cold Atmospheric Plasma Combined With Endovascular Intervention for Diabetic Foot Ulcers With Lower Extremity Arterial Occlusion: A Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: Efficacy and Safety of Cold Atmospheric Plasma Combined With Endovascular Intervention for Diabetic Foot Ulcers With Lower Extremity Arterial Occlusion
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shenyang Medical College (Other)
Collaborators: Ansteel Group General Hospital (Unknown)
Responsible Party: Principal Investigator, Lin Tao, Assoc. Prof., Shenyang Medical College
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAP_Foot_Ulcers
Record Dates: First submitted 2025-09-25; First posted 2025-09-30 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Diabetic Foot Ulcers (DFU); Lower Extremity Arterial Occlusion
Keywords: Cold Atmospheric Plasma; Diabetic Foot Ulcers; lower extremity arterial occlusion
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Intervention Model Description: This is a two-arm, parallel-assignment, randomized controlled trial. Participants are randomly assigned in a 1:1 ratio to receive either cold atmospheric plasma (CAP) therapy or sham CAP therapy, in addition to standard diabetic foot ulcer care. Both groups receive 10 treatment sessions over 10 consecutive days. The trial includes blinded outcome assessment and sham control procedures to preserve participant blinding.
Who Masked: Participant, Outcomes Assessor
Masking Description: To preserve procedural blinding, participants in the placebo group will undergo a simulated intervention using an identical device setup, with the plasma-generating electric field disabled. The system will mimic the treatment session environment (including operating sounds and airflow) without producing active plasma or gas.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cold Atmospheric Plasma (CAP) Group (Experimental): Participants with diabetic foot ulcers (DFUs) and infrapopliteal arterial occlusion who receive CAP therapy once daily for 10 days following successful endovascular intervention.
  Interventions: Device: Cold Atmospheric Plasma (CAP); Procedure: Infrapopliteal Endovascular Revascularisation; Other: Guideline-Based Standard DFU Care
- Sham CAP (Placebo) Group (Placebo Comparator): Participants with DFUs and infrapopliteal arterial occlusion who receive sham CAP therapy with an identical-looking device that does not produce active plasma.
  Interventions: Device: Sham CAP Therapy; Procedure: Infrapopliteal Endovascular Revascularisation; Other: Guideline-Based Standard DFU Care

INTERVENTIONS:
Device: Cold Atmospheric Plasma (CAP) — CAP-activated gas treatment developed by Xi'an Jiaotong University (Chinese patent No. ZL202110209052.X); administered once daily for 10 days, 25 minutes per session.
  Arms: Cold Atmospheric Plasma (CAP) Group
Device: Sham CAP Therapy — Identical equipment without plasma activation; simulates treatment environment (sound, airflow) for participant blinding.
  Arms: Sham CAP (Placebo) Group
Procedure: Infrapopliteal Endovascular Revascularisation — Balloon angioplasty is performed on infrapopliteal arteries with significant stenosis or occlusion. Technical success is defined as <30% residual stenosis, confirmed intraoperatively by digital subtraction angiography (DSA). Only patients with successful revascularisation are eligible for randomisation.
Other: Guideline-Based Standard DFU Care — All participants will receive diabetic foot ulcer (DFU) care according to current international and Chinese clinical guidelines

SUMMARY:
The goal of this clinical trial is to evaluate whether cold atmospheric plasma (CAP) combined with endovascular intervention can accelerate wound healing and improve safety outcomes in patients aged 18 to 80 years with diabetic foot ulcers (DFUs) complicated by lower extremity arterial occlusion.

The main questions it aims to answer are:

1. Does CAP treatment lead to a greater reduction in ulcer area by Week 4 compared to placebo?;
2. Is CAP therapy safe and well-tolerated in patients with DFUs after successful infrapopliteal revascularisation?;

Researchers will compare CAP treatment plus standard care to sham CAP (placebo) plus standard care to see if CAP improves wound healing more effectively and reduces adverse local symptoms.

Participants will:

1. Receive either active CAP therapy or sham CAP therapy once daily for 10 days following endovascular revascularisation
2. Undergo daily wound assessments for ulcer area, signs of infection, and pain scores
3. Complete quality-of-life questionnaires (EQ-5D and SF-12) at baseline and Week 4
4. Be followed through Week 4 to assess efficacy and safety endpoints

DETAILED DESCRIPTION:
Diabetic foot ulcers (DFUs) complicated by lower extremity arterial occlusion are difficult to heal, even after successful endovascular revascularisation, due to persistent microcirculatory impairment and chronic inflammation. Cold atmospheric plasma (CAP) has shown promising effects in promoting wound healing through antimicrobial activity, angiogenesis induction, and modulation of inflammatory responses. However, its efficacy and safety in the clinical treatment of DFUs remain to be validated in randomized controlled trials.

This prospective, randomized, placebo-controlled, single-center clinical trial aims to assess the efficacy and safety of CAP therapy, delivered as CAP-activated gas, in patients with DFUs who have undergone successful infrapopliteal balloon angioplasty. Participants will receive either active or sham CAP therapy once daily for 10 days, in addition to standard DFU care. The primary endpoint is the percentage reduction in ulcer area at Week 4. Secondary outcomes include time to early healing response, pain scores, quality of life, and local adverse events.

The results of this study are expected to provide clinical evidence supporting the use of CAP as an adjunctive therapy in ischemic diabetic foot wound management.

ELIGIBILITY:
Inclusion Criteria:

* 1)Age between 18 and 80 years; diagnosed with type 1 or type 2 diabetes mellitus; with HbA1c ≤10%;
* 2)Presence of at least one chronic foot ulcer persisting for ≥3 weeks, with no signs of healing despite guideline-directed standard care; ulcer classified as Wagner-Armstrong grade 1D or 2D;
* 3)Imaging-confirmed infrapopliteal arterial stenosis or occlusion, assessed by vascular ultrasound and/or computed tomography angiography (CTA); all patients must have undergone infrapopliteal balloon angioplasty, with successful target vessel revascularisation confirmed intraoperatively (≤30% residual stenosis);
* 4)Signed written informed consent prior to study participation.

Exclusion Criteria:

* 1)Concurrent use of negative pressure wound therapy (NPWT) or maggot debridement therapy;
* 2)Undergoing dialysis for end-stage renal disease;
* 3)Use of topical antibiotics with known biological activity on the wound;
* 4)Use of platelet-rich fibrin (PRF) for wound treatment;
* 5)Women of childbearing potential without effective contraception, or currently breastfeeding;
* 6)Presence of severe comorbidities involving other organ systems, with an estimated life expectancy of less than 6 months;
* 7)Participation in another clinical trial within the past 3 months, or currently enrolled in another clinical study;
* 8)Any condition deemed unsuitable for trial participation at the discretion of the investigators.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-10-09 (Actual); Primary Completion 2026-03-20 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Change in ulcer area (cm²) | assessed at baseline, Day 1 to Day 10 post-randomisation, and at Week 4
  Ulcer area will be measured at baseline, daily from Day 1 to Day 10, and at Week 4 post-randomisation. Measurements are obtained from calibrated wound photographs and analysed using ImageJ software. Primary endpoint will be analysed using a linear mixed-effects model to evaluate differences between groups over time.

SECONDARY OUTCOMES:
Time to 10% reduction in ulcer area | From baseline through Day 10 and Week 4 post-randomisation
  The time (in days) from baseline to the first documentation of ≥10% reduction in ulcer surface area compared to baseline, as measured by calibrated wound photography analysed using ImageJ software. Ulcer size is measured daily from Day 1 to Day 10 and at Week 4.
Mean change in pain score measured by Visual Analogue Scale (VAS) | Baseline; daily from Day 1 to Day 10; and at Week 4 post-randomisation
  Pain severity will be assessed using the 10-point Visual Analogue Scale (VAS), where 0 indicates no pain and 10 indicates the worst pain imaginable. Measurements will be taken at baseline, daily from Day 1 to Day 10, and at Week 4 post-randomisation. Change in VAS score over time will be compared between groups.
Change in quality of life (EQ-5D) | Baseline and Week 4 post-randomisation
  Health-related quality of life will be assessed using the EuroQol 5-Dimension 5-Level questionnaire (EQ-5D-5L) at baseline and Week 4 post-randomisation. The EQ-5D-5L descriptive system evaluates five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, each scored on a 5-point ordinal scale (1 = no problems, 5 = extreme problems).
Change in quality of life (SF-12) | Baseline and Week 4 post-randomisation
  Quality of life will be assessed using the 12-Item Short Form Health Survey (SF-12) at baseline and Week 4 post-randomisation. The SF-12 is a validated instrument designed to evaluate health-related quality of life across physical and mental health domains. It yields two composite summary scores: the Physical Component Summary (PCS) and the Mental Component Summary (MCS).
  Each component score typically ranges from 0 to 100, with higher scores indicating better health status.

OTHER OUTCOMES:
Incidence of skin irritation | Daily from baseline to Day 10 and at Week 4 post-randomisation
  The presence or absence of skin irritation at the treatment site will be recorded by trained clinical staff during each treatment session (Day 1-10) and at Week 4. Skin irritation includes erythema, rash, itching, or other subjective symptoms reported by the participant or observed by the investigator.
Incidence of local bleeding | Daily from baseline to Day 10 and at Week 4 post-randomisation
  Bleeding at the wound or treatment site will be assessed by visual inspection and clinical documentation. Events are recorded as present or absent at each time point, and severity (mild, moderate, severe) will be noted if applicable.
Incidence of local burning sensation | Daily from baseline to Day 10 and at Week 4 post-randomisation
  Participants will be asked to report any burning sensation at the treatment site during or after CAP exposure. Events will be recorded as present or absent, and graded based on severity. This outcome will help assess the tolerability of CAP treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Yun-En Liu, MD, Study Chair — Shenyang Medical College; Lin Tao, MM, Principal Investigator — Shenyang Medical College
Locations (1):
- Ansteel Group General Hospital, Anshan, Liaoning, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol